CLINICAL TRIAL: NCT00177060
Title: Topical Hydromorphone for Wound Healing
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No funding available.
Sponsor: Hordinsky, Maria K., MD (Individual)
Organization: University of Minnesota (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 0308M50994
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2010-03-01 (Estimated); Status verified 2010-02

CONDITIONS: Wound Healing
MeSH Terms: interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: hydromorphone

SUMMARY:
The hypothesis is that topical opioids will hasten wound healing in humans.

DETAILED DESCRIPTION:
This is based on our published data that morphine is a powerful stimulant of angiogenesis and our preclinical study of wounds in rats which demonstrate that topical opioids (morphine, hydromorphone and fentanyl) hasten healing of punch biopsy wounds. This study will focus on hydromorphone which was more powerful than morphine as a wound-healer in the rat study.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as normal, healthy volunteers age 18-65.

Exclusion Criteria:

* Known bleeding disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2003-10; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Healing rates and microvessel density will be compared statistically for the control-ointment versus hydromorphone-ointment subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hordinsky, MD, Principal Investigator — University of Minnesota; Robert Hebbel, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States